CLINICAL TRIAL: NCT02713802
Title: An Open-Label, Randomized, Two-Way Crossover Pilot Study of the Bioequivalence of Cudafol(R) and Diprivan(R) IV Administered as Single Intravenous Doses in Healthy Subjects
Brief Title: Pilot Study of Bioequivalence of Cudafol(R) and Diprivan(R) Administered as Single Intravenous Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cuda Anesthetics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CUDA-C2015-001
Record Dates: First submitted 2016-01-15; First posted 2016-03-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test product (Experimental): Propofol solution (1% [10 mg/mL]), via intravenous injection
  Interventions: Drug: Cudafol(R) (propofol, 1% [10 mg/mL])
- Reference product (Active Comparator): Propofol emulsion (1% [10 mg/mL]), via intravenous injection
  Interventions: Drug: Diprivan(R) (propofol, 1% [10 mg/mL])

INTERVENTIONS:
Drug: Cudafol(R) (propofol, 1% [10 mg/mL]) — Test product Cudafol(R) to be administered via 1 mg/kg bolus injection, then continuous infusion at 50 ug/kg/min for 15 minutes
  Arms: Test product
Drug: Diprivan(R) (propofol, 1% [10 mg/mL]) — Reference product Diprivan(R) to be administered via 1 mg/kg bolus injection, then continuous infusion at 50 ug/kg/min for 15 minutes
  Arms: Reference product

SUMMARY:
Evaluate pharmacokinetic/pharmacodynamic equivalence and safety and tolerability of single doses of Cudafol(R) and Diprivan(R) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese men and women, 18 to 55 years of age inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening. Females of child-bearing potential must be using an approved contraceptive method.

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* History or presence of clinically significant abnormal 12-lead electrocardiogram (ECG), blood pressure, or heart rate.
* Pregnant or nursing (lactating) women.
* Known hypersensitivity or allergy to propofol (or components of either formulation, including eggs, soybean oil or betadex sulfobutyl ether sodium) or any other forms of anesthesia, or has had a reaction to anesthesia in the past.
* Family history of malignant hyperthermia.
* History of drug or alcohol abuse (or tests positive at screening) or current smoker.
* Poor venous access in either arm.
* Tests positive for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antibody.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on pharmacokinetic parameter: Area Under Curve | 0-24 hours post dose
Bioequivalence based on pharmacokinetic parameter: Cmax | 0-24 hours post dose

SECONDARY OUTCOMES:
Pharmacokinetic parameter: Tmax | 0-24 hours post dose
Incidence of adverse events and tolerability | 7 days post dose
  Number of adverse events and local tolerability

IPD SHARING:
Plan to Share IPD: No